## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | A double-blind (sponsor unblind), randomized, placebo controlled, single and repeat escalating dose study to investigate the safety, tolerability, and pharmacokinetics of CCI15106 inhalation powder in healthy participants and participants with moderate chronic obstructive pulmonary disease (COPD) including evaluation of environmental and healthy by-stander exposure levels during dosing. |
| <b>Compound Number</b> | : | CCI15106 |
| <b>Effective Date</b> | · | 30-Oct-2018 |

# **Description:**

- The purpose of this RAP is to describe the planned safety, tolerability and pharmacokinetic analyses and outputs to be presented in the Clinical Study Report for the study 205822. This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.
- Bystander and Environmental Exposure Analyses is tabulated and reported in a separate report.

## **RAP Author(s):**

| Approver | | Date | Approval Method |
|----------|-------------------------|-------------|-----------------|
| PPD | Clinical Statistics, ID | 30-Oct-2018 | PharmaTMF |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD Evacutive Medical Director D&D Infectious | 29-Oct-2018 | Email Approval |
| Executive Medical Director, R&D Infectious Diseases | 29 <b>-</b> 001-2018 | Email Approval |
| PPD | 30-Oct-2018 | Email Approval |
| Director, Clinical Pharmacology | 30 001 2010 | Eman Approva |
| PPD | 29-Oct-2018 | PharmaTMF |
| Regional Study Manager, NLD CRT PCPS | 2) 001 2010 | T Harma Tivii |
| PPD | 29-Oct-2018 | PharmaTMF |
| Principal Clinical Data Manager, RD, PCPS | 29-OCI-2018 | Filatilia i IVII |
| PPD | 30-Oct-2018 | PharmaTMF |
| Associate Manager (ID, Clinical Programming) | 30-OCI-2018 | r IIai IIIa i Ivir |
| PPD | 29-Oct-2018 | PharmaTMF |
| Principal Programmer/Analyst, RD PCPS | 29 <b>-001-</b> 2018 | F Hallila I IVIF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|----------------------------------------------|-------------|-----------------|
| Statistics Director, RD PCPS | 30-Oct-2018 | PharmaTMF |
| Associate Manager (ID, Clinical Programming) | 29-Oct-2018 | PharmaTMF |

# **TABLE OF CONTENTS**

| 1. INTRODUCTION | 5 |
|---|---|
| 2.1. Changes to the Protocol Defined Statistical Analysis Plan 2.2. Study Objective(s) and Endpoint(s) 2.3. Study Design 2.4. Statistical Hypotheses 3. PLANNED ANALYSES 3.1. Interim Analyses 3.2. Final Analyses 4. ANALYSIS POPULATIONS 4.1. Protocol Deviations 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 5.1. Study Treatment & Sub-group Display Descriptors 5.2. Baseline Definitions 5.2.1. Baseline Definitions 5.2.2. Derivations and Handling of Missing Baseline Data 5.3. Other Considerations for Data Analyses and Data Handling | |
| 2.1. Changes to the Protocol Defined Statistical Analysis Plan 2.2. Study Objective(s) and Endpoint(s) 2.3. Study Design 2.4. Statistical Hypotheses 3. PLANNED ANALYSES 3.1. Interim Analyses 3.2. Final Analyses 4. ANALYSIS POPULATIONS 4.1. Protocol Deviations 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 5.1. Study Treatment & Sub-group Display Descriptors 5.2. Baseline Definitions 5.2.1. Baseline Definitions 5.2.2. Derivations and Handling of Missing Baseline Data 5.3. Other Considerations for Data Analyses and Data Handling | 5 |
| 2.2. Study Objective(s) and Endpoint(s). 2.3. Study Design | |
| 2.3. Study Design | |
| 2.4. Statistical Hypotheses | |
| 3.1. Interim Analyses 3.2. Final Analyses 4. ANALYSIS POPULATIONS 4.1. Protocol Deviations 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 5.1. Study Treatment & Sub-group Display Descriptors 5.2. Baseline Definitions 5.2.1. Baseline Definitions 5.2.2. Derivations and Handling of Missing Baseline Data 5.3. Other Considerations for Data Analyses and Data Handling | |
| 3.2. Final Analyses | 9 |
| 4. ANALYSIS POPULATIONS 4.1. Protocol Deviations 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 5.1. Study Treatment & Sub-group Display Descriptors 5.2. Baseline Definitions 5.2.1. Baseline Definitions 5.2.2. Derivations and Handling of Missing Baseline Data 5.3. Other Considerations for Data Analyses and Data Handling | |
| Protocol Deviations | 9 |
| 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS | |
| CONVENTIONS 5.1. Study Treatment & Sub-group Display Descriptors 5.2. Baseline Definitions 5.2.1. Baseline Definitions 5.2.2. Derivations and Handling of Missing Baseline Data 5.3. Other Considerations for Data Analyses and Data Handling | 10 |
| 5.2. Baseline Definitions | |
| 5.2.1. Baseline Definitions | 11 |
| <ul><li>5.2.2. Derivations and Handling of Missing Baseline Data</li><li>5.3. Other Considerations for Data Analyses and Data Handling</li></ul> | |
| 5.3. Other Considerations for Data Analyses and Data Handling | |
| 6. STUDY POPULATION ANALYSES | |
| 6.1. Overview of Planned Study Population Analyses | |
| 6.1.1. Disposition and Withdrawals | |
| 6.1.2. Demographic and other Baseline Characteristics | |
| 6.1.3. Medications | |
| 7. SAFETY ANALYSES | 16 |
| 7.1. Study Medication Exposure | |
| 7.2. Adverse Events Analyses | 17 |
| 7.3. Clinical Laboratory Analyses | 18 |
| 7.4. ECG Evaluations | |
| 7.5. Telemetry Evaluations | |
| 7.6. Spirometry Evaluations | |
| 7.7. Vital Signs | |
| 7.8. Bystander and Environmental Exposure Analyses | 19 |
| 8. PHARMACOKINETIC ANALYSES | |
| 8.1. Overview of Planned Pharmacokinetic Analyses | |
| 8.1.1. Drug Concentration Measures | 20 |
| 8.1.1.1. Derivation of Lung ELF Drug (CCI15106) Concentration Data | 24 |
| 8.1.2. Pharmacokinetic Parameters | |
| 8.1.2.1. Deriving Pharmacokinetic Parameters | |

## CONFIDENTIAL

| | | | 8.1.2.2. | Statistical Analysis of Pharmacokinetic Parameters | 23 |
|---|---|---|---|---|---|
| 9. | POPU | LATION F | PHARMACO | OKINETIC (POPPK) ANALYSES | 24 |
| 10. | REFE | RENCES. | | | 25 |
| 11. | | | | | 26 |
| | 11.1. | | | ol Deviation Management and Definitions for Per | |
| | | Protocol | Population | | 26 |
| | 44.0 | | | s from Per Protocol Population | |
| | 11.2. | | | ule of Activities | |
| | 44.0 | | | Defined Schedule of Events | 27 |
| | 11.3. | | | Phases and Treatment Emergent Adverse | 22 |
| | | 11.3.1. | | ases | |
| | | 11.5.1. | | Study Phases for Concomitant Medication | |
| | | 11.3.2. | | t States for Adverse Events Data | |
| | 11.4. | | | isplay Standards & Handling Conventions | |
| | 11.7. | 11.4.1. | | Process | |
| | | 11.4.2. | | Standards | |
| | | 11.4.2. | | Standards for Pharmacokinetic | |
| | 11.5. | _ | | d and Transformed Data | |
| | 11.5. | 11.5.1. | | d and Transionned Data | |
| | | 11.5.1. | | oulation | |
| | | 11.5.3. | | | |
| | 11.6. | | | ing Standards for Missing Data | |
| | 11.0. | 11.6.1. | | e Withdrawals | |
| | | 11.6.2. | | of Missing Data | |
| | | 11.0.2. | | Handling of Missing and Partial Dates | |
| | 11.7. | Annendix | 7. Values | of Potential Clinical Importance | 39 |
| | | | | y Values | |
| | | 11.7.2. | , | , | |
| | | | | S | |
| | 11.8. | | | C Dataset Specification | |
| | 11.9. | | | riations & Trade Marks | |
| | | | | ions | |
| | | | | ks | |
| | 11.10. | | | f Data Displays | |
| | | | | lay Numbering | |
| | | | | mple Shell Referencing | |
| | | | | les | |
| | | 11.10.4. | Study Pop | oulation Tables | 46 |
| | | 11.10.5. | Safety Tak | bles | 50 |
| | | 11.10.6. | Pharmaco | okinetic Tables | 57 |
| | | | | okinetic Figures | |
| | | | | gs | |
| | | | | Listings | |
| | 11.11. | | | ple Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology | | |
|---------------------|-------------|-------------|
| 2016N290366_02 | 11-OCT-2017 | Amendment 2 |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Bystander and Environmental Exposure Analyses will be reported in a separate report.

The Lung ELF Concentration population for analysis is renamed to BAL PK in order to keep it consistent with the other Phase I study (202031).

The All Participants Screened, Safety, Systemic Pharmacokinetic Concentration (PK), the BAL PK analysis populations are not defined separately for Part 1 and Part 2 as mentioned in the protocol.

For the data disclosure outputs regarding "Summary of Age Ranges", the Enrolled population is defined in this RAP.

The term "Subjects" is used to refer to the "Participants" in certain sections of this document including the TFLs.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | | Endpoints | |
|---|---|---|---|
| Pri | Primary Objectives | | Primary Endpoints |
| • | To investigate the safety and tolerability of CCI15106-IP following single and repeat escalating doses in healthy participants and participants with moderate COPD. | • | Adverse events (AEs), clinical laboratory, electrocardiogram (ECG), telemetry, spirometry, and vital signs assessments. |
| • | To determine systemic PK of CCI15106 following single and repeat escalating doses of CCI15106-IP in healthy participants and participants with moderate COPD. | • | Derived systemic PK parameters of CCI15106: Single dose: area under the curve (AUC) from time zero to the time of last quantifiable concentration (AUC[0-last]), concentration at maximum (Cmax), time of maximum concentration (tmax), AUC from time zero to infinity (AUC[0- $\infty$ ]) elimination half-life (t1/2), clearance (CL/F), as data permit. Repeat dose: AUC from time zero to end of dosing interval (AUC[0- $\tau$ ]) ( $\tau$ =12 hours [h] for twice daily dose regimen), Cmax, tmax, elimination half-life (t1/2) as data permit. |
| • | To evaluate potential inhalation exposure of bystanders to airborne | • | Concentration of CCI15106 in plasma of bystanders 15-<br>20 minutes (min) after dosing (at predicted tmax) and |

| Objectives | Endpoints |
|---|---|
| CCI15106 during self-administered dosing of participants. | amount of CCI15106 accumulated on filters fitted on bystander over 15 min after dosing. |
| To evaluate the distribution and persistence of airborne CCI15106 in room air post-dosing. | Amount of CC15106 in room air assessed by measuring amount of CC115106 accumulated over 20 and 60 min intervals during and immediately post-dosing on filters fitted on stationary pumps placed in the room. |
| Secondary Objectives | Secondary Endpoints |
| To determine the concentration of<br>CCI15106 in the lung of healthy<br>participants and participants with<br>moderate COPD following repeat<br>dosing of CCI15106-IP. | Concentrations of CCI15106 in lung epithelial lining fluid (ELF) assessed by bronchoalveolar lavage (BAL). |
| To investigate the performance of the<br>Monodose RS01 device for the<br>administration of CCI15106-IP in<br>healthy participants and participants<br>with moderate COPD. | Device safety and performance parameters, including<br>medical device incidents reporting, as well as systemic<br>PK and lung CCI15106 concentrations. |
| Exploratory Objectives | Exploratory Endpoints |
| To assess dose proportionality of<br>CCI15106-IP versus systemic PK<br>parameters. | <ul> <li>Comparisons of doses administered and systemic PK<br/>parameters of CCI15106: AUC(0-24) or AUC(0-τ) and<br/>Cmax.</li> </ul> |
| To explore the relationship of drug exposure to safety and tolerability parameters after single and repeat escalating doses of CCI15106-IP in healthy participants and participants with moderate COPD. | The dose or plasma exposure parameters for CCI15106 and the relationship of these to safety and tolerability parameters, as data permit. |
| To extrapolate study outcomes to a<br>realistic worst case real-life scenario<br>of dosing multiple patients in a single<br>room in a nursing home. | Comparison of the study room with a potential nursing<br>home room, including room dimensions, patient density,<br>ventilation (air change rates per hour). |

## 2.3. Study Design





# 2.4. Statistical Hypotheses

The primary objective of the study is to investigate the safety and tolerability of CCI15106-IP following single and repeat escalating doses in healthy participants and participants with moderate COPD. No statistical hypotheses will be tested.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal interim analyses are planned for this study. Safety and tolerability will be evaluated as described in Section 2.3. Systemic and, where available, lung PK may also be evaluated.

# 3.2. Final Analyses

Safety and PK analyses are the primary statistical analyses for this study.

Data will be listed and summarized according to GSK reporting standards, where applicable. All the displays will be split by part. Study population tables would be presented by cohort and a combined placebo (of all cohorts with the exception of Part 1, Cohort C (bystanders)). For Safety displays, listings will be sorted by dose, participant and time; summaries will be presented by dose and time for different parts of the study. Participants receiving placebo may be combined into one treatment group in the summaries within each part.

Descriptive summaries will include n, mean, standard deviation (SD), median, minimum, and maximum, geometric mean with associated 95% confidence interval (CI), and the between-participant coefficient of variation (%CVb) for continuous variables related to PK parameters, n and percent will be used as summary statistics for categorical variables.

Version 9.4 or higher of the SAS system will be used to analyse the data as well as to generate tables, figures, and listings.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Screened | Comprises of all participants who consent to participate in the clinical study. | Screen Failures |
| Enrolled | <ul> <li>All participants who passed screening and entered the study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| Safety | <ul> <li>Comprises of all participants who receive at least one dose of study treatment during the study.</li> <li>This population will be based on the treatment the participant actually received.</li> </ul> | <ul><li>Safety</li><li>Study Population</li></ul> |
| Systemic<br>Pharmacokinetic<br>Concentration<br>(PK) | <ul> <li>Participants who receive at least one dose of study treatment and who undergo plasma PK sampling and have at least one post-dose concentration result.</li> <li>PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether</li> </ul> | • PK |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | or not the sample will be excluded. | |
| BAL PK | Healthy participants who receive at least one dose of<br>study treatment and who undergo BAL sampling and<br>have post-dose lung ELF CCI15106 and urea<br>concentration result. | • BAL |
| | Lung ELF samples that may be affected by protocol deviations, will be reviewed by the study team to determine whether or not the sample will be excluded. | |
| Bystander Safety | Participants who are present at least once in the room | Safety |
| Population (Part 1, Cohort C) | with the participant receiving the dose. | Study Population |
| Bystander PK<br>Population (Part<br>1, Cohort C) | Participants who are present at least once in the room with the participant receiving the dose, undergo plasma PK sampling and have post-dose concentration result. | • PK |
| | PK samples that may be affected by protocol deviations<br>will be reviewed by the study team to determine whether<br>or not the sample will be excluded. | |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.

 This dataset will be the basis for the summaries and listings of protocol deviations.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned examinations of covariates and subgroups.
- There are no planned adjustments made for multiple centres in this study as this is a single centre study.
- There are no planned adjustments for multiple comparisons or multiplicity.

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | | |
|---|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | | |
| Code | Description | Display Header | Footnote Treatment<br>Description | Order [1] |
| S1 | CCI15106-IP 60<br>mg – Single Dose | CCI15106 SD 60mg(HV) | CCI15106-IP 60 mg<br>Single Dose for Part 1,<br>Cohort A | 1 |
| S2 | CCI15106-IP 120<br>mg – Single Dose | CCI15106 SD 120mg(HV) | CCI15106-IP 120 mg<br>Single Dose for Part 1,<br>Cohort A | 2 |
| R1 | CCI15106-IP 30<br>mg - BID | CCI15106 BID 30mg(HV) | CCI15106-IP 30 mg BID for Part 1, Cohort A | 3 |
| R2 | CCI15106-IP 60<br>mg - BID | CCI15106 BID 60mg(HV) | CCI15106-IP 60 mg BID<br>For Part 1, Cohort B | 4 |
| Р | Placebo | Placebo(HV) | Placebo for Part 1 Cohorts<br>A and B | 5 |
| S1 | CCI15106-IP 60<br>mg – Single Dose | CCI15106 SD<br>60mg(COPD) | CCI15106-IP 60 mg<br>Single Dose for Part 2,<br>Cohort A COPD | 6 |
| R2 | CCI15106-IP 60<br>mg - BID | CCI15106 BID<br>60mg(COPD) | CCI15106-IP 60 mg BID for Part 2, Cohort B COPD | 7 |
| Р | Placebo | Placebo(COPD) | Placebo for Single Dose and BID for COPD | 8 |
| BYS | Bystander Cohort | Bystander | Bystander | 9 |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

## 5.2. Baseline Definitions

#### 5.2.1. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

For tabulated safety summaries, only the scheduled assessments will be included in the summary tables.

| Parameter | Study Assessn | Study Assessments Considered as Baseline | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-<br>Dose) | in Data Display |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | - | Х | Day 1 (Pre-Dose) |
| Spirometry | Х | - | X | Day 1 (Pre-Dose) |
| Haematology/Chemistry/Urinalysis | Х | X | - | Day - 1 |
| Telemetry | - | - | X | Day 1 (Pre-Dose) |

#### NOTES:

 Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

## 5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.2.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data are missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on change from baseline displays wherever applicable.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.2 | Appendix 2: Assessment Windows |
| 11.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |

## CONFIDENTIAL

## 

| Section | Component |
|---------|-----------------------------------------------------|
| 11.6 | Appendix 6: Reporting Standards for Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

All the displays will be split by part. Study population tables would be presented by cohort and a combined placebo (of all cohorts).

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomization | | | |
| Randomization | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | Υ | | Υ |
| Reason for Screening Failures | Y | | Υ |
| Reason for Withdrawals | | | Υ |
| Protocol Deviations | Y | | Υ |
| Inclusion and Exclusion Criteria Deviations | | | Υ |
| Study Populations | Υ | | |
| Demography | | | |
| Demographics Characteristics | Υ | | Υ |
| Race & Racial Combinations | Y | | Υ |
| Medical Condition & Concomitant Medications | | | |
| Medical Conditions (Current/Past) | Y | | Υ |
| Concomitant Medications | Y | | Y |

#### NOTES:

# **6.1.1.** Disposition and Withdrawals

All participants who provide informed consent will be accounted for in this study. In each study part, subject disposition will be tabulated for each study treatment and for all participants combined with the number of participants who are randomly assigned to treatment, complete the study and prematurely discontinue as well as the reason for early discontinuation. A listing will present dates of completion or early withdrawal and the reason for early discontinuation, if applicable, for each participant.

Listings of study eligibility, treatment randomization and study treatment administration will be provided for each study part based on the layout mentioned above.

<sup>•</sup> Y = Yes display generated.

## 6.1.2. Demographic and other Baseline Characteristics

Individual subject demographics and baseline characteristics (medical history and results from drug and alcohol screens, smoking/nicotine history) will be presented in listings for each study part.

Demographic characteristics such as age, sex, race, ethnicity, height, weight, and body mass index (BMI) will be summarized and tabulated by treatment and for all participants overall for each study part. Descriptive statistics will be presented for age, height, weight, and BMI. Frequency counts and percent will be presented for sex, race and ethnicity.

#### 6.1.3. Medications

All prior and concomitant medications will be listed for each study part based on the layout mentioned earlier. Summaries of all medications taken during the course of the study will be presented in tabular form for each study part using GSK Drug Dictionary 1.3. The number and percentage of participants taking concomitant medications will be summarized by cohort and overall for each study part separately. For each participant, the medication will be counted only once within a given preferred drug name level. A participant may appear more than once if he/she has more than one concomitant medication coded under different categories, however, the participant will be counted only once in the overall category.

Please refer to Appendix 3: Study Phases and Treatment Emergent Adverse Events for definition of prior, concomitant and post-treatment medications. Handling of partial dates for medications is outlined in Appendix 6: Reporting Standards for Missing Data.

## 7. SAFETY ANALYSES

The primary safety analyses for this study will be based on the Safety population for each dose taken, analysed separately for study parts, unless otherwise specified.

Data will be listed and summarized according to GSK reporting standards, where applicable. Listings will be sorted by dose, participant and time; summaries will be presented by dose and time for different parts of the study. Participants receiving placebo may be combined into one treatment group in the summaries within each part.

For categorical variables, the population size (N for sample size and n for available data) and the percentage (of available data) for each class of variable will be presented. Continuous variables will be summarized using descriptive statistics, including N, mean, standard deviation (SD), median, minimum and maximum values.

Table 3 provides an overview of the planned safety analyses for each study part, unless otherwise specified, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| Endpoint | | Abs | olute | | ( | Change fro | m Baselin | ie |
|---|---|---|---|---|---|---|---|---|
| | Summary | | | ridual | Sum | mary | | ridual |
| | T | F | F | L | T | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | Υ | | | Υ | | | | |
| Adverse Events <sup>1</sup> | | | | | | | | |
| All AE's | Υ | | | Υ | | | | |
| Serious AE's | Υ | | | Υ | | | | |
| Treatment related AE's | Υ | | | Υ | | | | |
| AE's leading to | Υ | | | Υ | | | | |
| Withdrawal | | | | | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry <sup>2</sup> | Υ | | | Υ | Υ | | | |
| Hematology | Υ | | | Υ | Υ | | | |
| Coagulation | Υ | | | Υ | | | | |
| Urinalysis | | | | Υ | | | | Υ |
| ECG's <sup>3</sup> | | | | | | | | |
| ECG Findings | Υ | | | Υ | | | | |
| ECG Values | Υ | | | Υ | Υ | | | |
| Vital Signs <sup>3</sup> | | | | | | | | |
| Vitals Values | Υ | | | Υ | Υ | | | |
| Spirometry | | | | | | | | |
| Spiromtery | Υ | | | Υ | | | | |
| Telemetry | | | | | | | | |
| Telemetry Findings | Υ | | - | Υ | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Listings will include participant's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text.
- 2. Chemistry summaries will include both changes from baseline & emergent results by PCI criteria.
- 3. Listings and summaries for ECGs and vital signs include treatment emergent PCI results

# 7.1. Study Medication Exposure

Exposure to study medication as the number of doses administered will be presented for each treatment for each Part.

# 7.2. Adverse Events Analyses

Adverse Events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, Version 21.0.

See Appendix 3: Study Phases and Treatment Emergent Adverse Events to determine treatment states for AE data. Handling of partial dates for AEs is outlined in Appendix 6: Reporting Standards for Missing Data. In the rare case when it is not possible to assess treatment emergence, the AE will be classified as treatment emergent (i.e. the worst case).

AE Severity is classified as mild (grade = 1), moderate (grade = 2), or severe (grade = 3). AEs with a missing severity will be classified as severe. If a participant reports an AE more than once within that SOC (System Organ Class)/ PT (Preferred Term), the AE with the worst case severity will be used in the corresponding severity summaries.

Relationship to study treatment, as indicated by the Investigator, is classified as "not related" or "related". AEs with a missing relationship to study medication will be regarded as "related" to study medication.

All AE tabulations will be performed separately for Part 1 and Part 2, by dose, and will include the number and percentage of participants. For each study part and cohort, incidence of AEs will be tabulated by the following:

- All AEs by SOC and PT
- All related AEs by SOC and PT
- All AEs by SOC, PT and Severity
- All related AEs by SOC, PT and Severity

All AEs leading to permanent discontinuation of study treatment will be identified by using the variable pertaining to outcome on the Adverse Events page of the CRF, and listed separately for each study part and cohort.

Serious adverse events (SAEs) are those events recorded as "Serious" on the Adverse Events page of the CRF, and will be listed separately for each study part.

The details of the planned displays are provided in Appendix 11: List of Data Displays.

# 7.3. Clinical Laboratory Analyses

Laboratory results will be included in the reporting of this study for hematology, coagulation, clinical chemistry, and urinalysis.

Protocol-specified clinical laboratory tests will be summarized using descriptive statistics. The statistics will be presented for each scheduled assessment during the study and change from baseline to each scheduled assessment. Presentations will use SI Units, as provided by the labs or converted from values in other units. Clinical laboratory data collected during unscheduled visits of study conduct that were not required per protocol, such as for special testing to evaluate an AE, will be listed and not summarized.

Based upon laboratory normal ranges, the laboratory test results will be categorized according to the normal range as low (below the lower limit), normal (within the normal range) and high (above the upper limit). Summary statistics for change from baseline based on PCI will also be tabulated. The details of the planned displays are in Appendix 11: List of Data Displays.

## 7.4. ECG Evaluations

The following ECG parameters will be reported for each study part: PR, QRS, QT, QTc, QTcF and HR (bpm). Replicate quantitative values taken per time point will be averaged for all analysis and reporting. Summary statistics for change from baseline will also be tabulated.

Overall assessment of ECG (Investigator's judgment) will be recorded as follows:

- Normal
- Abnormal, Not Clinically Significant
- Abnormal, Clinically Significant

# 7.5. Telemetry Evaluations

Overall assessment of Telemetry (Investigator's judgment) will be recorded as follows:

Normal

- Abnormal, Not Clinically Significant
- Abnormal, Clinically Significant

All measurements will be listed.

# 7.6. Spirometry Evaluations

The following parameters will be reported for each timepoint: FEV1 and FVC. The maximum of the measurements will be calculated. All measurements will be listed.

% Predicted Normal FEV1 = (Max FEV1/Predicted Normal FEV1)x100

% Predicted FVC = (Max FVC/Predicted Normal FVC)x100

# 7.7. Vital Signs

The following Vital Signs measurements will be reported for each study part: supine systolic and diastolic blood pressure, pulse rate, respiratory rate and temperature.

For participants undergoing BAL, vital signs will also include oxygen saturation.

Triplicate quantitative values taken per time point will be averaged for all analysis and reporting.

Summary statistics for collected vital signs, change from baseline, and summary of PCI will also be tabulated.

# 7.8. Bystander and Environmental Exposure Analyses

The bystander and environmental analysis will be analyzed and presented in a separate report.

## 8. PHARMACOKINETIC ANALYSES

# 8.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the "Systemic Pharmacokinetic Concentration" population for the plasma drug concentration data, and "BAL PK Population" for the lung ELF concentration data, unless otherwise specified.

Table 4 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Pharmacokinetic Analyses

| Endpoints | | | Untr | ransfo | rmed | | | | | Log-1 | ransf | ormed | ł | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | Summary | | Individual | | Stats Analysis | | | mary | Individual | |
| | T | F | L | T | F | F | L | Т | F | Ш | Т | F | F | L |
| Plasma Drug<br>Concentrations | | | | Y | Y [1] [2] [3] [4] | Y<br>[1] | Υ | | | | | Y<br>[1]<br>[2] | Y<br>[1] | |
| Derived PK<br>Parameters | Υ | | | Υ | | | Υ | Υ | Y<br>[7] | Y<br>[8] | | | | |
| Lung ELF CCI15106<br>Concentration | | | | Υ | <b>Y</b><br>[5] | <b>Y</b><br>[6] | Υ | | | | | | Y<br>[1] | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (± SD) and Median plots will be generated, for the BD cohorts, overlay the day 1 and day 14 on same plot where possible.
- 3. Mean (± SD) and Median plots by cohorts a) to compare over the first 12hours for 60mg in HV (part 1) and COPD (part 2); b) to compare the 60mg SD (over 24h) HV vs COPD; c) to compare the 60mg BD HV vs COPD one for each of the intense sampling day (day 1, day 14).
- 4. Boxplot of plasma drug concentration at the follow up visit by cohort.
- 5. Boxplot of Lung CCI15106 concentration by cohort (HV vs COPD).
- 6. Lung CCI15106 concentration by Subject ID.
- 7. Dose proportionality of single and repeat dose and accumulation ratios from Cohorts A and B will be evaluated in Part 1 and Part 2.
- 8. Supportive SAS Output from Statistical Analysis of Loge-transformed Plasma PK Parameters.

## 8.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions.

## 8.1.1.1. Derivation of Lung ELF Drug (CCI15106) Concentration Data

Urea concentration data will be used to calculate the dilution effect of the BAL A correction for dilution will be applied to all BAL drug concentrations as follows:

$$Lung\ Drug\ Concentration(ng/mL) = \frac{BAL}{Drug\ Concentration}(ng/mL) \times DilutionFactor$$

where

$$Dilution\ Factor = \frac{Plasma\ Urea_{pre-BAL}}{BAL\ Urea}$$

#### 8.1.2. Pharmacokinetic Parameters

## 8.1.2.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions for the treatment of concentrations below the assay's lower limit of quantification (LLQ).
- The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin<sup>™</sup> 6.4 or higher (Pharsight Corporation, a Certara Company, Princeton, NJ), and/or SAS<sup>™</sup> Version 9.4 or higher. Graphics may be prepared using the same versions of SAS<sup>™</sup>, or Phoenix WinNonlin<sup>™</sup>, or with SigmaPlot<sup>™</sup> 12.5, or higher (Systat Software, Inc., San Jose, California).
- All calculations of non-compartmental parameters will be based on actual sampling times, except for the purpose of interim reviews where nominal sampling times will be used.
- Pharmacokinetic parameters described in Table 5 (Cohorts A, Part 1 and Part 2) and Table 6 (Cohort A, Part 1, Cohorts B, Part 1 and Part 2) will be determined from the plasma concentration-time data, as data permits, for CCI15106 (ribavirin).

Table 5 Derived Pharmacokinetic Parameters (Cohorts A, Part 1 and Part 2 – Single dose)

| Parameter | Parameter Description |
|---|---|
| AUC <sub>(0-t)</sub> | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (ng·h/mL) after each single dose will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC <sub>(0-∞)</sub> | Area under the concentration-time curve extrapolated to infinity (ng·h/mL) will be calculated by linear up/log down trapezoidal summation as: |
| | $AUC = AUC_{(0-t)} + C(t) / \lambda_z$ |
| AUC <sub>(0-12)</sub> | Area under the concentration-time curve from time zero to 12 hours post dose, e.g. for |

| Parameter | Parameter Description |
|---|---|
| | cohort A part 1, AUC <sub>(0-12)</sub> will be calculated after the 60mg SD (day 1), 120mg SD (day 3), and first dose of 30mg BD (day 6) |
| AUC <sub>(0-24)</sub> | Area under the concentration-time curve from time zero to 24 hours post dose, e.g. for cohort A part 1, AUC <sub>(0-24)</sub> will be calculated after the 60mg SD (day 1), 120mg SD (day 3) |
| AUC <sub>(0-48)</sub> | Area under the concentration-time curve from time zero to 48 hours post dose, e.g. for cohort A part 1, AUC <sub>(0-24)</sub> will be calculated after the 60mg SD (day 1), 120mg SD (day 3) |
| C <sub>max</sub> | Maximum observed concentration in plasma (ng/mL), determined directly from the concentration-time data. |
| t <sub>max</sub> | Time to reach C <sub>max</sub> (h), determined directly from the concentration-time data. |
| t <sub>1/2</sub> | Apparent terminal half-life (h) will be calculated as: $t_{1/2} = \ln 2 / \lambda_z$ |
| $\lambda_z$ | Apparent terminal rate constant (1/h), determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points will be used for determination. |
| CL/F | Apparent inhaled plasma clearance after dosing (L/h), calculated as administered dose divided by $AUC(0-\infty)$ . |

#### NOTES:

Additional parameters may be included as required.

Table 6 Derived Pharmacokinetic Parameters (Cohort A, Part 1, Cohorts B, Part 1 and Part 2 – Repeat Dose)

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the concentration-time curve in the plasma during a dosing interval (ng·h/mL) on day 1 and day 14, calculated by linear up/log down trapezoidal summation. Actual elapsed time at the end of the dosing interval will be used for the calculation. $\tau$ =12 for BID dosing regimen |
| C <sub>max</sub> | Maximum observed concentration in plasma (ng/mL), determined directly from the concentration-time data. |
| t <sub>max</sub> | Time to reach C <sub>max</sub> (h), determined directly from the concentration-time data. |
| t <sub>1/2</sub> | Apparent terminal half-life (h) will be calculated as:<br>$t_{1/2} = \ln 2 / \lambda_z$ |
| $\lambda_z$ | Apparent terminal rate constant (1/h), determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points will be used for determination. |

#### NOTES:

Additional parameters may be included as required.

Individual lung ELF concentration data will be summarised, listed and displayed graphically on both linear and semi-logarithmic scales for the Cohorts with available ELF data. Where data permit, the individual lung ELF concentration data may be plotted against the plasma concentration measured prior to BAL sampling.

## 8.1.2.2. Statistical Analysis of Pharmacokinetic Parameters

Geometric mean will be included for PK parameters, wherever applicable.

The following PK statistical analyses will only be performed, if sufficient data is available (i.e. if participants have well defined plasma profiles).

## Pharmacokinetic Statistical Analyses

#### Endpoint(s)

- All endpoints, except tmax and %AUCex, will be natural-log transformed prior to the analysis
- Dose Proportionality: AUC<sub>(0-24)</sub> or AUC<sub>(0-48)</sub>, or AUC<sub>(0-τ)</sub> and Cmax, for single dose and repeat dose of Part 1
- Steady State Assessment in BID dosing: Ctrough (using pre-dose concentration from day 6 in Cohort A Part 1, and day 2 onwards in Cohorts B, Part 1 and Part 2)
- Accumulation in BID dosing: accumulation ratio will be calculated for AUC<sub>(0-τ)</sub> as [AUC<sub>(0-τ)</sub>, on Day 19/AUC<sub>(0-τ)</sub>, on Day 6 for Cohort A in Part 1, or AUC<sub>(0-τ)</sub> on Day 14/AUC<sub>(0-τ)</sub> on Day 1 for Cohorts B of both Part 1 and Part 2, from the ANOVA model

#### Model Specification

Dose Proportionality will be assessed separately by means of power model: y = α\*dose<sup>β</sup> where y
denotes the PK parameter being analyzed. PK parameters will be normalized to 60mg dose and then
log transformed prior to analysis

If the power model does not show dose proportionality then pairwise analysis of variance (ANOVA) may be used as an exploratory analysis to understand the dose where dose proportionality fails

- Analysis of variance (ANOVA), considering study Day as fixed effect and subject as a random effect in
  the model, will be performed using SAS Mixed Linear Models procedure to evaluate in the assessment
  of steady state in models included at least 3 days of pre-dose concentrations (like Days 4,6,8; Days
  6,8,10, Days 10,12,14 relative to first dose of repeat dosing). This will be done for each of the repeat
  dose treatments.
- Analysis of variance (ANOVA), considering study Day as fixed effect and subject as a random effect in
  the model, will be performed using SAS Mixed Linear Models procedure to evaluate in the assessment
  accumulation, where geometric least squares mean ratio of AUC<sub>(0-τ)</sub> on Day 19/AUC<sub>(0-τ)</sub> on Day 6 for
  Cohort A in Part 1, AUC<sub>(0-τ)</sub> on Day 14/AUC<sub>(0-τ)</sub> on Day 1 for Cohorts B and 90% CI will be calculated.

Note: Subjects will be fit as a fixed effect for the assessment of accumulation if the model fails to converge.

Estimates of within-subject variability for Cmax, t1/2, AUC<sub>(0-r)</sub> and CL/F will be provided, where CVw(%) = SQRT(exp(MSE) – 1)×100 and MSE is the residual mean squared error from the model. CVw represents a pooled measure of within-subject variability in repeat dose group.

#### Model Results Presentation

- Dose Proportionality: The intercept α and the slope β with corresponding 90% CIs will be estimated and presented for each PK parameter
- Steady State Assessment: Estimated slope parameter with 90% CI will be presented.
- Accumulation and Time Invariance: Geometric means with 90% CIs by parameter and day will be
  presented. Ratio of geometric means with corresponding 90% CIs for Day 14/ Day 1 for Cohort B or
  Day 19/Day 6 for Cohort A of Part 1 will also be presented.
- Comparative Plot of Individual Plasma PK Parameter Versus Treatment will be generated.
- Individual and box plots of Pre-dose concentrations will be generated.
- The SAS output from the statistical models will be included in a listing of supportive SAS output.

# 9. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Population pharmacokinetics modelling may be conducted and reported separately.

The detailed PopPK methodology will be described in a separate RAP where appropriate. The required data for the analyses are provided in Appendix 8: Population Pharmacokinetic (PopPK) Analyses and are subject to delivery soon after DBF.

# 10. REFERENCES

GlaxoSmithKline Document Numbers 2015N238595\_00 (Original – 24-SEP-2015): A Double-Blind, Placebo-Controlled, Dose Escalation, First Time in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of GSK3389404 in Healthy Subjects.

Whitehead J. Easy-to-implement Bayesian methods for dose-escalation studies in healthy subjects. *Biostatistics*. 2001; 2:47-61.

- 11. APPENDICES
- 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population
- 11.1.1. Exclusions from Per Protocol Population

N/A

# 11.2. Appendix 2: Schedule of Activities

# 11.2.1. Protocol Defined Schedule of Events

# Screening and follow-up procedures for all cohorts

| Procedure | Screening, ≤ 30<br>days before D1 for<br>Part 1 or ≤ 45 days<br>before D1 for Part<br>21 | Follow up<br>30±2 days after the<br>last dosing day | Notes |
|---|---|---|---|
| Informed consent | Х | | Screening assessments can be performed over multiple screening visits |
| Inclusion and exclusion criteria | X | | <ol><li>If test otherwise performed within 3 months prior to first dose of study treatment, testing</li></ol> |
| Demography | X | | at screening is not required |
| Full physical examination including<br>height and weight, oral examination | Х | | To be drawn fasting (for at least 8 h) To be administered to participants with COPD only, 15-30 minutes prior to spirometry |
| Brief physical examination, oral examination | | Х | To be done at screening for participants with COPD only, following salbutamol dosing To be performed in the bronchoalveolar lavage (BAL) cohorts only to confirm participant |
| Medical history (includes substance<br>usage and Family history of<br>premature CV disease) | х | | eligibility 7. To be performed in the BAL cohorts only to confirm participant eligibility. Can be done pre-dose on Day -1 instead, if required |
| Substance testing (drugs, alcohol) | X | | |
| Assessment of child-bearing potential<br>for females | Х | | |
| Serum pregnancy test in women | X | X | |
| Human immunodeficiency virus (HIV),<br>Hepatitis B (Hep B) and Hepatitis C<br>(Hep C) screen <sup>2</sup> | Х | | |
| Haematology, clinical chemistry and<br>urinalysis (include liver chemistries) <sup>3</sup> | Х | X | |
| Salbutamol administration <sup>4</sup> | X | | |
| Spirometry <sup>5</sup> | X | | |
| 12-lead ECG and vital signs | Х | X | |
| Coagulation parameters6 | X | | |
| Capillary pCO <sub>2</sub> <sup>7</sup> | X | | |
| PK blood sample | | X | |
| AE review | | X | |
| SAE review | X | X | |
| Concomitant medication review | Х | X | |

## Schedule for Cohort A Part 1

| Procedure | | | | | | | | | | Tre | atmer | nt Peri | od, Da | ys | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | 11 | 2 | 31 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 |
| Inclusion and exclusion criteria | Х | | | | | | | | | | | | | | | | | | | | | | |
| Brief physical examination, oral examination | Χ | | | | | | | | | | | | | | | | | | | | | | Х |
| Substance testing (drugs, alcohol, tobacco) | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Inhaler device training <sup>2</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Serum pregnancy test in women | X | | | | | | | | | | | | | | | | | | | | | | |
| Admittance to clinic | X | | | | | | | | | | | | | | | | | | | | | | |
| Randomization | X3 | | | | | | | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | | | | | | | X4 |
| Haematology, clinical chem and urinalysis (include liver chem) <sup>5</sup> | Χ | | X | | | χ | | | | | | | Χ | | | | | | | | | | Х |
| Spirometry | | X1 | | X1 | | | Х6 | | <b>X</b> <sup>7</sup> | | | X <sup>7</sup> | | | | | X7 | | | Χ6 | | | |
| Telemetry (starting 30 min pre-morning dose and continuous at least 4h post-morning dose) | | X1 | | X1 | | | Х | | | | | | Х | | | | | | Х | | | | |
| 12-lead ECG and vital signs | XX | Χ¹ | | Χ¹ | | | X8 | | X8 | X8 | | X8 | X8 | X8 | | X8 | | X8 | | | | | |
| CCI15106-IP or placebo treatment, device incident assessment | | X1 | | X1 | | | X9 | X <sup>9</sup> | X9 | X <sup>9</sup> | X9 | X9 | X9 | X9 | X9 | X9 | X9 | X9 | X <sup>9</sup> | X9 | | | |
| PK blood sample <sup>10</sup> | | Х | Х | Χ | Х | Х | Х | Х | | Χ | | Х | | Х | | Х | | Х | | Х | Х | Χ | X |
| AE review | | | <del>(-==</del> | | | | | | | | | | | | | | | | | | | <del>-</del> | |
| SAE review | | <del>(</del> | | | | | | | | | | | | | | | | | | | | <del>)</del> | |
| Concomitant medication review | | <del>(</del> === | | | | | | | | | | | | | | | | | | | | <del>-</del> | |

- 1. Single dose days. Follow schedule for Day 1 of Part 2 Cohort A
- 2. Day -1 inhaler training may be done on Day 1 instead, before the first dose administration. Other time-points may be added per investigators discretion.
- 3. Can be performed on Day 1 prior to dosing
- 4. After all procedures and assessments are complete
- 5. To be drawn fasting (for at least 8 h)
- 6. To be performed at the following timepoints in the mornings only: pre-dose, and 0.25, 0.5, 1, 4 h post-dose
- 7. To be performed at the following timepoints in the mornings only: pre-dose and 4 h post-dose
- 8. ECG and vital signs to be obtained 2 h after the morning dose
- BI
- 10. PK samples on days 1, 3, 6, and 19 will be collected at the following timepoints: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 h. On day 2, one sample in the morning (24h post day 1 dose). On days 4 and 5, one sample on each morning (24h and 48h post day 3 dose). On days 6 and 19, the evening dose will be given after 12 h post-dose sample is collected. On all other days, PK sample will be collected once, before the morning dose (if on dosing days).

# Schedule for Cohort A Part 2 (and all other single dose administrations)

| | Treatment Period, Days (D) and hours (h) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | D-1 D1 | | | | | | | | | | | | | D2 |
| Procedure | | Pre-<br>dose | 0h | 0.25h | 0.5h | 0.75h | 1h | 2h | 4h | 6h | 8h | 10h | 12h | 24h |
| Inclusion and exclusion criteria | X | | | | | | | | | | | | | |
| Brief physical examination, oral examination | X | | | | | | | | | | | | | Х |
| Substance testing (drugs, alcohol) | X | | | | | | | | | | | | | |
| Serum pregnancy test in women | X | | | | | | | | | | | | | |
| Admittance to clinic | X | | | | | | | | | | | | | |
| Inhaler device training <sup>1</sup> | Х | | | | | | | | | | | | | |
| Randomization | X2 | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | Х3 |
| Haematology, clinical chem and urinalysis (include liver chem)4 | Χ | | | | | | | | | | | | | Χ |
| Spirometry | | X5 | | X6 | Χ | | Χ6 | | Х6 | | | | | |
| Telemetry | | 30 min pre-dose and continuous until at least 4 h | | | | | | | | | | | | |
| 12-lead ECG and vital signs | | XXX | | X | | | Χ | X | X | | Χ | | Χ | |
| CCI15106-IP or placebo treatment | | | Х | | | | | | | | | | | |
| PK blood sample <sup>7</sup> | | Х | | Х | X | X | Х | Х | Х | Χ | Х | Х | X | Х |
| AE review | ←→ | | | | | | | | | | | | | |
| SAE review | <del>(</del> | | | | | | | | | | | | | |
| Concomitant medication review | <del>(</del> ====== | | | | | | | | | | | | | <del>-</del> |

- 1. Day -1 inhaler training may be done on Day 1 instead, before the first dose administration. Other time-points may be added per investigators discretion
- 2. Can be performed on Day 1 prior to dosing
- 3. After all assessments are completed
- 4. To be drawn fasting (for at least 8 h)
- 5. To be performed within 15 to 60 minutes pre-dose
- 6. To be performed after ECG, VS and PK blood draw are obtained
- 7. Additional PK collection time points may be added to better characterize the PK profile

# Repeat dose schedule to be followed for repeat dose cohorts in Parts 1 and 2 (other than Cohort A Part 1)

| Procedure | | | | | | | Trea | tment P | eriod, [ | Days | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Inclusion and exclusion criteria | X | | | | | | | | | | | | | | | |
| Brief physical examination, oral examination | X | | | | | | | | | | | | | | | X |
| Substance testing (drugs, alcohol, tobacco1) | X | | | | | | | | | | | | | | | |
| Inhaler device training <sup>2</sup> | X | | | | | | | | | | | | | | | |
| Serum pregnancy test in women | X | | | | | | | | | | | | | | | |
| Admittance to clinic | X | | | | | | | | | | | | | | ĺ | |
| Randomization | X <sub>3</sub> | | | | | | | | | | | | | | 1 | |
| Discharge | | | | | | | | | | | | | | | ĺ | X4 |
| Dosing procedure training with bystanders | | χ5 | | | | | | | | | | | | | 1 | |
| Haematology, clinical chem and urinalysis (include liver chem)6 | Х | | | | | | | Х | | | | | | | | Х |
| Spirometry | | <b>X</b> 7 | | Χ8 | | | Χ8 | | | | | Χ8 | | | Х7 | |
| Telemetry (starting 30 min pre-morning dose and continuous at least 4h post-morning dose) | | Х | | | | | | Х | | | | | | X <sup>9</sup> | | |
| 12-lead ECG and vital signs <sup>10</sup> | XXX | Χ | | Χ | Χ | | Х | Х | Χ | | X11 | | X11 | | ĺ | |
| CCI15106-IP or placebo treatment BID, device incident assessment BID <sup>12</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| PK blood sample <sup>13</sup> | | Χ | Х | | Χ | | Х | | Χ | | Х | | Х | | Х | X |
| BAL | | | | | | | | | | | X14 | | | | | |
| Urea blood sample | χ15 | | | | | | | | | | | | | | | |
| AE review | ( | | | | | | | | | | | | | | | |
| SAE review | <del>(</del> | | | | | | | | | | | | | | | |
| Concomitant medication review | <del>(</del> | | | | | | | | | | | | | | | <del>&gt;</del> |

- 1. Tobacco test to be performed only in healthy participants
- 2. Day -1 inhaler training may be done on Day 1 instead, before the first dose administration. Other time-points may be added per investigators discretion.
- 3. Can be performed on Day 1 prior to dosing
- 4. After all procedures and assessments are complete
- 5. To be done only in Cohort(s) where bystanders are present. Can be performed on Day -1 instead, if desired. Other time-points may be added per investigators discretion.
- 6. To be drawn fasting (for at least 8 h)
- 7. To be performed at the following timepoints in the mornings only: pre-dose, and 0.25 (in participants with COPD only), 0.5, 1, 4 h post-dose
- 8. To be performed at the following timepoints in the mornings only: pre-dose and 4 h post-dose

- 9. Telemetry may be performed on Days 11 or 12 instead, not to coincide with the BAL procedure.
- 10. ECG and vital signs to be obtained 2 h after the morning dose
- 11. When BAL is performed, vital signs and ECG will be performed before and after the procedure and oxygen saturation will be measured continuously.
- 12. For cohort with bystanders, BID doses may have ±1.5 h window.
- 13. PK samples on days 1 and 14 will be collected at the following timepoints: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 h. The evening dose will be given after 12 h post-dose sample is collected. On all other days, PK sample will be collected once, before the morning dose. When BAL is performed, one additional PK sample will be collected after dosing immediately prior to bronchoscopy
- 14. Done once during these four days, as soon as possible (within 1 h) after the first dose of the day
- 15. To be collected immediately before bronchoscopy

## Schedule for Cohort C Part 1 (bystanders and air monitoring), to be executed concomitantly with Cohort B Part 1

| Procedure Treatment Period, Days | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Inclusion and exclusion criteria | Х | | | | | | | | | | | | | | | |
| Brief physical examination, oral examination | Х | | | | | | | | | | | | | | | Х |
| Substance testing (drugs, alcohol, tobacco) | X | | | | | | | | | | | | | | ĺ | |
| Serum pregnancy test in women | X | | | | | | | | | | | | | | | |
| Admittance to clinic | X | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | X1 |
| Training <sup>2</sup> | X | | | | | | | | | | | | | | | |
| Haematology, clinical chem and urinalysis (include liver chem)3 | X | | | | | | | Χ | | | | | | | | Χ |
| Exposure to dosing | | Χ | Χ | X | X | X | X | Χ | Χ | X | Χ | X | X | X | Χ | |
| PK blood sample | | X <sup>4</sup> | | | | | | X <sup>4</sup> | | | | | | | X <sup>4</sup> | X |
| Stationary pump air monitoring <sup>5</sup> | | Χ | | | | | | Χ | | | | | | | Χ | |
| Personal exposure pump monitoring <sup>6</sup> | | Χ | | | | | | Χ | | | | | | | Χ | |
| 12-lead ECG and vital signs | XXX | X7 | | <b>X</b> <sup>7</sup> | <b>X</b> <sup>7</sup> | | X7 | <b>X</b> <sup>7</sup> | X7 | | <b>X</b> <sup>7</sup> | | <b>X</b> <sup>7</sup> | | | |
| AE review | <b>←</b> | | | | | | | | | | | | | | | |
| SAE review | ← | | | | | = <del>-&gt;</del> | | | | | | | | | | |
| Concomitant medication review | <del>(</del> | | | | | | = <del>-&gt;</del> | | | | | | | | | |

- 1. After all procedures and assessments are complete
- 2. Day -1 training may be done on Day 1 instead, before the first dose administration. Other time-points may be added per investigators discretion
- 3. To be drawn fasting (for at least 8 h)
- 4. PK samples will be collected pre-dose and 15 min after the dosing participant takes their first daily dose. In addition, on days 7 and 14, one sample on each day will be collected before the dosing participant takes the first daily dose. On day 15, one sample will be collected before discharge.
- 5. Samples of air to be collected for 20 and 60 min during and after the first morning dose
- 6. Samples of air to be collected for 15 min during and after the first morning dose
- 7. ECG and vital signs to be obtained 2 h after the exposure to morning dose

# 11.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 11.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

# 11.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 11.3.2. Treatment States for Adverse Events Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date if AE start time not available; else |
| Pre-rreatment | AE Start Date time < Study Treatment Start Date time |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date |
| Since 1st Dose | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |
| (Days) | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF OR value is missing. |

# NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

# 11.4.1. Reporting Process

#### Software

 The currently supported versions of SAS software will be used to perform all data analyses, generate tables, figures and listings.

# **Reporting Area**

| HARP Server | : us1salx00259 |
|---------------|---------------------------------------|
| HARP Compound | : \arprod\cci15106\mid205822\final_03 |

# Analysis Datasets

- Analysis datasets will be created according to CDISC standards (AdaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files may be generated for SAC tables...

## 11.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the CRF.
- The reported precision from non CRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits</li> </ul> | Unscheduled visits will not be included in summary tables. |
| <ul> <li>Unscheduled visits</li> </ul> | Unscheduled visits will not be included in figures. |
| All unscheduled vis | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. and Standards for the Transfer and Reporting of PK Data using HARP | |

# 11.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Insert document name]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Parameter Data | |
| Descriptive Summary<br>Statistics (Log<br>Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log-transformed data and between geometric coefficient of variation (CVb (%)) will be reported.<br>[1] $CV_b$ (%) = $\sqrt{\exp(SD^2) - 1}$ * 100 (SD = SD of log transformed data) |
| Parameters Not<br>Being Log<br>Transformed | N, n, geometric mean, 95% CI (Lower, Upper), standard deviation (SD), median, minimum and maximum |
| Listings | Interval, number of observations included in calculation of lambda_z, regression coefficient and percent AUC extrapolated (%AUCex) |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety
  parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of
  related summary tables. This will also be applicable to relevant Potential Clinical Importance summary
  tables.

## **Study Day**

- Calculated as the number of days from randomisation date:
  - Ref Date = Missing
    - → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Date ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

# 11.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

## **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

## Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

## **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
### 11.5.3. Safety

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1

Example 3: 0 Significant Digits = '< x' becomes x - 1

## 11.6. Appendix 6: Reporting Standards for Missing Data

### 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all visits of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data are not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data are excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 11.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.7. Appendix 7: Values of Potential Clinical Importance

## 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Con | cern Range |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | ~/I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |
| [Insert as Required] | [Units] | | | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|----------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |

### 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Abaaluta OTa Intamial | | > 450 | <480 |
| Absolute QTc Interval | msec | ≥ 480 | < 500 |
| | | ≥ 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 [ | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 30 | < 60 |
| | msec | ≥ 60 | |

# 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|----------|
| (Change from Baseline) | | Decrease | Increase |
| Systolic Blood Pressure | mmHg | ≥ 40 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 20 | ≥ 20 |
| Heart Rate | bpm | ≥ 30 | ≥ 30 |

## 11.8. Appendix 8: Pop PK Dataset Specification

For the purpose of population PK analysis, the raw plasma concentration data in the systemic PK population (including all the available plasma concentration data) will be merged for each individual with the following demographic and baseline/screening variables where available. In addition, the 12-ECG data as listed below will be merged with plasma concentration data by the planned time.

The dataset will be a comma delimited ASCII text file, named as: NM.205822.PK.v1.csv.

| Variable | Description | Format | Unit | Missing | Note |
|---|---|---|---|---|---|
| AGE | Subject Age | Num | Specify | -99 | From source data. |
| SEX | Subject gender | Integer | None | Never | 0=Male, 1=Female |
| SEXTEXT | Subject gender text | Char | None | Never | Text corresponding to code for SEX |
| BMI | Baseline Body<br>Mass Index | Num | Specify | -99 | From source data. Formula: Weight(kg)/(height(m)**2) |
| WT | Baseline Subject weight | Num | Specify | -99 | From source data. |
| HT | Baseline Subject height | Num | Specify | -99 | From source data. |
| RACE | Subject race code1 | Integer | None | -99 | From source data e.g. 1=African American / African Heritage 2=American Indian or Alaska Native 3=Asian – Central / South Asian Heritage 4=Asian – East Asian Heritage 5=Asian – Japanese Heritage 6=Asian – South East Asian Heritage 7=Asian – Mixed Race 8=Native Hawaiian or other Pacific Islander 9=White – Arabic / North African Heritage 10=White – White / Caucasian / European Heritage 11=White – Mixed Race 12=Mixed Race |
| RACETXT | Subject race text | Char | None | Never | Text corresponding to code for RACE |
| ETHN | Subject ethnicity | Num | None | -99 | From source data definition. E.g 1=Hispanic or Latino, 2=Non-Hispanic |
| ETHNTEXT | Subject ethnicity text | Char | None | Never | Text corresponding to code for ETHN. |
| SCR | Serum Creatinine | Num | micromol/L | -99 | Baseline/screening defined in the source dataset |
| CRCL | Baseline<br>Creatinine<br>Clearance | Num | mL/min | -99 | From source data. formula e.g. Creatinine Clearance will be calculated based on the Cockcroft-Gault equation. • CrCL (ml/min) = [140 – AGE (in years)]*Weight(kg)*0.85 (for female patients) / [72* Serum Creatinine (micromol/L) * 0.0113 |
| ALT | Alanine aminotransferase | Num | | -99 | Baseline/screening defined in the source dataset |
| AST | Aspartate aminotransferase | Num | | -99 | Baseline/screening defined in the source dataset |
| ALB | Albumin | Num | | -99 | Baseline/screening defined in the source |

| Variable | Description | Format | Unit | Missing | Note |
|---|---|---|---|---|---|
| | | | | | dataset |
| TBIL | Total bilirubin | Num | | -99 | Baseline/screening defined in the source dataset |
| ECGTM | Clock time of ECG recording in hours | Num | | | ECGTM should be calculated as: hr + min/60 e.g. if clock time of ECG recording is 09:30, then ECGTM= 9 + 30/60= 9.5 |
| HR | Heart rate in bpm | Num | bpm | | As in source dataset |
| HRBL | Baseline heart rate in bpm | Num | bpm | | As in source dataset |
| PR | PR interval in ms | Num | ms | | As in source dataset |
| PRBL | Baseline<br>corresponding PR<br>interval in ms | Num | ms | | As in source dataset |
| QRS | QRS complex duration in ms | Num | ms | | As in source dataset |
| QRSBL | Baseline<br>corresponding<br>QRS interval in ms | Num | ms | | As in source dataset |
| QT | Uncorrected QT interval in ms | Num | ms | | As in source dataset |
| QTBL | Baseline<br>uncorrected QT<br>interval in ms | Num | ms | | As in source dataset |
| QTcF | QT with Fridericia's correction in ms | Num | ms | | As in source dataset |
| QTcFBL | Baseline QT with<br>Fridericia's<br>correction in ms | Num | ms | | As in source dataset |
| RR | RR interval in ms | Num | ms | | As in source dataset |
| RRBL | Baseline<br>corresponding RR<br>interval in ms | Num | ms | | As in source dataset |

# 11.9. Appendix 9: Abbreviations & Trade Marks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | |
| CDISC | Analysis and Reporting |
| CI | Clinical Data Interchange Standards Consortium Confidence Interval |
| CPMS | |
| | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QĊ | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| וטעט | Stady Data Standardization i lan |

| Abbreviation | Description |
|--------------|------------------------------|
| SDTM | Study Data Tabulation Model |
| SoA | Schedule of Activities |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ADVAIR |
| SAS |
| SigmaPlot |
| WinNonlin |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |

### 11.10. Appendix 10: List of Data Displays

### 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|-------------|
| Study Population | 1.1 to 1.30 | N/A |
| Efficacy | N/A | N/A |
| Safety | 3.1 to 3.60 | N/A |
| Pharmacokinetic | 4.1 to 4.7 | 4.1 to 4.12 |
| Population Pharmacokinetic (PopPK) | N/A | N/A |
| Pharmacodynamic and / or Biomarker | N/A | N/A |
| Pharmacokinetic / Pharmacodynamic | N/A | N/A |
| Section | List | ings |
| ICH Listings | 1 to | 66 |
| Other Listings | 66 to 82 | |

### 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|------------------------------------------------|
| DS [X] | During Study |
| DE [X] | Dose Escalation |
| IA SAC [X] | Interim Analysis Statistical Analysis Complete |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 11.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Participant Disposition – Part 1 | The general layout of all the study population tables would follow mock shell SAFE_T1 for the column headers and order for both Part 1 and Part 2 tables. | SAC |
| | | | | This will not include Cohort C, Part 1. | |
| 1.2. | Safety | ES1 | Summary of Participant Disposition – Part 2 | | SAC |
| 1.3. | Bystander<br>Safety (Part<br>1, Cohort C) | ES1 | Summary of Participant Disposition – Bystander | Only for Cohort C, Part 1. | SAC |
| 1.4. | All<br>Participants<br>Screened) | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.5. | All<br>Participants<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part 2 | | SAC |
| 1.6. | All<br>Participants<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure – Bystander | Only for Cohort C, Part 1. | SAC |
| Protoc | ol Deviation | | | | |
| 1.7. | Safety | DV1 | Summary of Important Protocol Deviations – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.8. | Safety | DV1 | Summary of Important Protocol Deviations – Part 2 | | SAC |

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | Bystander<br>Safety (Part<br>1, Cohort C) | DV1 | Summary of Important Protocol Deviations - Bystander | Only for Cohort C, Part 1. | SAC |
| Popula | tion Analysed | | | | • |
| 1.10. | All Screened | SP1A | Summary of Study Populations – Part 1 | | SAC |
| 1.11. | All Screened | SP1A | Summary of Study Populations – Part 2 | | SAC |
| 1.12. | Bystander<br>Safety (Part<br>1, Cohort C) | SP1A | Summary of Study Populations – Bystander | Only for Cohort C, Part 1. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | • | |
| 1.13. | Safety | DM1 | Summary of Demographic Characteristics – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.14. | Safety | DM1 | Summary of Demographic Characteristics – Part 2 | | SAC |
| 1.15. | Bystander<br>Safety (Part<br>1, Cohort C) | DM1 | Summary of Demographic Characteristics – Bystander | Only for Cohort C, Part 1. | SAC |
| 1.16. | Safety | DM5 | Summary of Race and Racial Combinations – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.17. | Safety (Part<br>2) | DM5 | Summary of Race and Racial Combinations – Part 2 | | SAC |
| 1.18. | Bystander<br>Safety (Part<br>1, Cohort C) | DM5 | Summary of Race and Racial Combinations – Bystander | Only for Cohort C, Part 1. | SAC |
| 1.19. | Safety | DM6 | Summary of Race and Racial Combination Details – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.20. | Safety (Part<br>2) | DM6 | Summary of Race and Racial Combination Details – Part 2 | | SAC |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.21. | Bystander<br>Safety (Part<br>1, Cohort C) | DM6 | Summary of Race and Racial Combination Details – Bystander | Only for Cohort C, Part 1. | SAC |
| 1.22. | Enrolled | DM11 | Summary of Age Ranges – Part 1 | This will not include Cohort C, Part 1. Please include the footnote: "[1] Age is calculated based on screening date, using date of birth, truncated to integer value. Note that only the year of birth has been collected where the day and month would be 30th June for all subjects." | SAC |
| 1.23. | Enrolled | DM11 | Summary of Age Ranges – Part 2 | Please include the footnote: "[1] Age is calculated based on screening date, using date of birth, truncated to integer value. Note that only the year of birth has been collected where the day and month would be 30th June for all subjects." | SAC |
| 1.24. | Enrolled | DM11 | Summary of Age Ranges – Bystander | Only for Cohort C, Part 1. Please include the footnote: "[1] Age is calculated based on screening date, using date of birth, truncated to integer value. Note that only the year of birth has been collected where the day and month would be 30th June for all subjects." | SAC |

| Study I | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 1.25. | Safety | MH1 | Summary of [Current/Past] Medical Conditions – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.26. | Safety | MH1 | Summary of [Current/Past] Medical Conditions – Part 2 | | SAC |
| 1.27. | Bystander<br>Safety (Part<br>1, Cohort C) | MH1 | Summary of [Current/Past] Medical Conditions - Bystander | Only for Cohort C, Part 1. | SAC |
| 1.28. | Safety | CM1 | Summary of Concomitant Medications – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.29. | Safety | CM1 | Summary of Concomitant Medications – Part 2 | | SAC |
| 1.30. | Bystander<br>Safety (Part<br>1, Cohort C) | CM1 | Summary of Concomitant Medications – Bystander | Only for Cohort C, Part 1. | SAC |
| 1.31. | Safety | NS1 | Summary of Number of Subjects by Country and Site ID - Part 1 | This will not include Cohort C, Part 1. | SAC |
| 1.32. | Safety | NS1 | Summary of Number of Subjects by Country and Site ID - Part 2 | | SAC |
| 1.33. | Bystander<br>Safety (Part<br>1, Cohort C) | NS1 | Summary of Number of Subjects by Country and Site ID -<br>Bystander | Only for Cohort C, Part 1. | SAC |

# 11.10.5. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term – Part 1 | The general layout of all the safety tables would follow mock shell SAFE_T4 for the column headers and order for both Part 1 and Part 2 tables. This will not include Cohort C, Part 1. | SAC |
| 3.2. | Safety | AE1 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term – Part 2 | | SAC |
| 3.3. | Bystander<br>Safety (Part<br>1, Cohort C) | AE1 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term – Bystander | | SAC |
| 3.4. | Safety | AE1 | Summary of Treatment Related Adverse Events by System Organ Class and Preferred Term – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.5. | Safety | AE1 | Summary of Treatment Related Adverse Events by System Organ Class and Preferred Term – Part 2 | | SAC |
| 3.6. | Bystander<br>Safety (Part<br>1, Cohort C) | AE1 | Summary of Treatment Related Adverse Events by System<br>Organ Class and Preferred Term – Bystander | | SAC |
| 3.7. | Safety | AE5A | Summary of Treatment Emergent Adverse Events by System Organ Class and Maximum Severity – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.8. | Safety | AE5A | Summary of Treatment Emergent Adverse Events by System Organ Class and Maximum Severity – Part 2 | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | Bystander<br>Safety (Part<br>1, Cohort C) | AE5A | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Maximum Severity – Bystander | | SAC |
| 3.10. | Safety | AE5A | Summary of Treatment Related Adverse Events by System Organ Class and Maximum Severity – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.11. | Safety | AE5A | Summary of Treatment Related Adverse Events by System<br>Organ Class and Maximum Severity – Part 2 | | SAC |
| 3.12. | Bystander<br>Safety (Part<br>1, Cohort C) | AE5A | Summary of Treatment Related Adverse Events by System<br>Organ Class and Maximum Severity – Bystander | | SAC |
| 3.13. | Safety | AE1 | Summary of All Serious Adverse Events – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.14. | Safety | AE1 | Summary of All Serious Adverse Events – Part 2 | | SAC |
| 3.15. | Bystander<br>Safety (Part<br>1, Cohort C) | AE1 | Summary of All Serious Adverse Events – Bystander | Only for Cohort C, Part 1. | SAC |
| 3.16. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.17. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study – Part 2 | | SAC |
| 3.18. | Bystander<br>Safety (Part<br>1, Cohort C) | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from the Study – Bystander | | SAC |
| Labora | tory: Chemistry | I | | | |
| 3.19. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.20. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit – Part 2 | | SAC |
| 3.21. | Bystander<br>Safety (Part<br>1, Cohort C) | LB1 | Summary of Chemistry Changes from Baseline by Visit –<br>Bystander | Only for Cohort C, Part 1. | SAC |
| 3.22. | Safety | LB17 | Summary of Clinical Chemistry Values by Potential Clinical Importance – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.23. | Safety | LB17 | Summary of Clinical Chemistry Values by Potential Clinical Importance – Part 2 | | SAC |
| 3.24. | Bystander<br>Safety (Part<br>1, Cohort C) | LB17 | Summary of Clinical Chemistry Values by Potential Clinical Importance – Bystander | Only for Cohort C, Part 1. | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.25. | Safety | LB1 | Summary of Haematology Changes from Baseline by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.26. | Safety | LB1 | Summary of Haematology Changes from Baseline by Visit – Part 2 | | SAC |
| 3.27. | Bystander<br>Safety (Part<br>1, Cohort C) | LB1 | Summary of Haematology Changes from Baseline by Visit – Bystander | Only for Cohort C, Part 1. | SAC |
| 3.28. | Safety | LB17 | Summary of Hematology Values by Potential Clinical Importance – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.29. | Safety | LB17 | Summary of Hematology Values by Potential Clinical Importance – Part 2 | | SAC |
| 3.30. | Bystander<br>Safety (Part<br>1, Cohort C) | LB17 | Summary of Hematology Values by Potential Clinical Importance – Bystander | Only for Cohort C, Part 1. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Coagulati | on | | | |
| 3.31. | Safety | LB1 | Summary of Coagulation Changes from Baseline by Visit – Part 1 | Only for Cohorts B, Part 1. | SAC |
| 3.32. | Safety | LB1 | Summary of Coagulation Changes from Baseline by Visit – Part 2 | Only for Cohorts B, Part 2. | SAC |
| Teleme | try | | | | |
| 3.33. | Safety | Non-standard<br>SAFE_T2 | Summary of Telemetry Findings – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.34. | Safety | Non-standard<br>SAFE_T2 | Summary of Telemetry Findings – Part 2 | | SAC |
| Spirom | etry | | | | |
| 3.35. | Safety | Non-standard<br>SAFE_T3 | Summary of Spirometry Data – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.36. | Safety | Non-standard<br>SAFE_T3 | Summary of Spirometry Data – Part 2 | | SAC |
| ECG | | | | | |
| 3.37. | Safety | EG1 | Summary of ECG Findings by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.38. | Safety | EG1 | Summary of ECG Findings by Visit – Part 2 | | SAC |
| 3.39. | Bystander<br>Safety (Part<br>1, Cohort C) | EG1 | Summary of ECG Findings by Visit – Bystander | Only for Cohort C, Part 1. | SAC |
| 3.40. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.41. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit – Part 2 | | SAC |
| 3.42. | Bystander<br>Safety (Part<br>1, Cohort C) | EG2 | Summary of Change from Baseline in ECG Values by Visit – Bystander | Only for Cohort C, Part 1. | SAC |
| 3.43. | Safety | Non-standard<br>SAFE_T7 | Frequency of Maximum ECG Values by PCI Category – Part 1 | Compute and display Maximum by day. | SAC |
| 3.44. | Safety | Non-standard<br>SAFE_T7 | Frequency of Maximum ECG Values by PCI Category – Part 2 | | SAC |
| 3.45. | Bystander<br>Safety (Part<br>1, Cohort C) | Non-standard<br>SAFE_T7 | Frequency of Maximum ECG Values by PCI Category – Bystander | Compute and display Maximum by day. Only for Cohort C, Part 1. | SAC |
| 3.46. | Safety | Non-standard<br>SAFE_T8 | Frequency of Worst Change from Baseline Values of QTcB and QTcF by PCI Category – Part 1 | Compute and display Maximum by day. | SAC |
| 3.47. | Safety | Non-standard<br>SAFE_T8 | Frequency of Worst Change from Baseline Values of QTcB and QTcF by PCI Category – Part 2 | | SAC |
| 3.48. | Bystander<br>Safety (Part<br>1, Cohort C) | Non-standard<br>SAFE_T8 | Frequency of Worst Change from Baseline Values of QTcB and QTcF by PCI Category – Bystander | Compute and display Maximum by day. Only for Cohort C, Part 1. | SAC |
| Vital Si | gns | | | | |
| 3.49. | Safety | VS1 | Summary of Vital Signs by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.50. | Safety | VS1 | Summary of Vital Signs by Visit – Part 2 | | SAC |
| 3.51. | Bystander<br>Safety (Part<br>1, Cohort C) | VS1 | Summary of Vital Signs by Visit – Bystander | Only for Cohort C, Part 1. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.52. | Safety | VS1 | Summary of Change from Baseline in Vital Signs by Visit – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.53. | Safety | VS1 | Summary of Change from Baseline in Vital Signs by Visit – Part 2 | | SAC |
| 3.54. | Bystander<br>Safety (Part<br>1, Cohort C) | VS1 | Summary of Change from Baseline in Vital Signs by Visit – Bystander | Only for Cohort C, Part 1. | SAC |
| 3.55. | Safety | VS2 | Summary of Vital Signs by PCI – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.56. | Safety | VS2 | Summary of Vital Signs by PCI – Part 2 | | SAC |
| 3.57. | Bystander<br>Safety (Part<br>1, Cohort C) | VS2 | Summary of Vital Signs by PCI - Bystander | Only for Cohort C, Part 1. | SAC |
| Exposu | re and Treatment | Compliance | | | |
| 3.58 | Safety | Non-standard<br>SAFE_T5 | Summary of Extent of Exposure to Study Treatment – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 3.59 | Safety | Non-standard<br>SAFE_T5 | Summary of Extent of Exposure to Study Treatment – Part 2 | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.60 | Bystander<br>Safety (Part<br>1, Cohort C) | Non-standard<br>SAFE_T5 | Summary of Extent of Exposure to Study Treatment – Bystander | | SAC |

## 11.10.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration Data | a | | | |
| 4.1. | Systemic PK | PK01 | Summary of CCI15106 Plasma Pharmacokinetic Concentration-<br>Time Data [ng/mL] by Cohort and Visit | | SAC |
| 4.2. | Systemic PK | PK01 | Summary of plasma CCI15106 Concentration Data at Follow Up visit [ng/mL] by Cohort | This will not include Cohort C, Part 1. | SAC |
| 4.3. | BAL PK | PK01 | Summary of Lung ELF CCI15106 Concentration Data [ng/mL] by Cohort | | SAC |
| PK Der | ived Parameter | S | | | |
| 4.4. | Systemic PK | PK03 | Summary of Derived CCI15106 Plasma Pharmacokinetic Parameters by Cohort and Visit | This will not include Cohort C, Part 1. | SAC |
| 4.5. | Systemic PK | Non-Standard<br>PK_T1 | Summary of Assessment of Dose Proportionality (Part 1 and Part 2) | Only for Cohorts A, Part 1 and Part 2. | SAC |
| 4.6. | Systemic PK | Non-Standard<br>PK_T2 | Summary of Assessment of Steady State (Part 1 and Part 2) | This will not include Cohort C, Part 1. | SAC |
| 4.7. | Systemic PK | Non-Standard<br>PK_T3 | Summary of Assessment of Accumulation (Part 1 and Part 2) | For Cohort A, Cohort B, Part 1, and Cohort B, Part 2. | SAC |

# 11.10.7. Pharmacokinetic Figures

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Mean/N | ledian Concent | tration Plots | | | |
| 4.1. | Systemic PK | PK17 | Mean (+SD) CCI15106 Plasma Concentration-Time Plot (Linear and Semi-log) (Part 1) | For Part 1, Overlay all cohorts and doses on same page, plot time upto 1) 72 hours post dose 2) 12 hours post dose [excluding the data after the 2 <sup>nd</sup> dose following the BD doses for both 1] & 2] to see better the earlier timepoitns. 3) plot to overlay day 1 and day 14 after the 30mg BD | SAC |
| 4.2. | Systemic PK | PK17 | Mean (+SD) CCI15106 Plasma Concentration-Time Plot (Linear and Semi-log) (Part 2) | For Part 2, 1) overlay day 1 and day 14 for each cohort (doses); 2) overlay all cohorts (doses) on same page for each full PK sampling day, Day 1 and Day 14 | SAC |
| 4.3. | Systemic PK | PK17 | Mean (+SD) CCI15106 Trough Plasma Concentration by study day (Linear and Semi-log) (Part 1 and Part 2) | Overlay the all cohorts on same page | SAC |
| 4.4. | Systemic PK | PK17 | Mean (+SD) CCI15106 Plasma Concentration-Time Plot by Cohort (to compare between HV and COPD) (Linear and Semilog) | 1) plot to overlay only data after 60mg SD (part 1 cohort A and part 2 cohort A) 2) plot to overlay data after 60mg BD (part 1 cohort B and part 2 cohort B), overlay all full PK sampling day (day 1 and day 14) as well as population on same page | SAC |
| 4.5. | Systemic PK | | Boxplot of pre-BAL plasma concentration by cohort (Linear and Semi-log) | Create a legend mentioning: Cohort B, Part 1 – Healthy Cohort B Part 2 - COPD | SAC |

| Pharm | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.6. | BAL PK | | Boxplot of Lung ELF CCI15106 concentration by cohort (Linear and Semi-log) | | SAC |
| Individ | ual Concentrati | on Plots | | | |
| 4.7. | Systemic PK | PK16a | Individual CCI15106 Plasma Concentration-Time Plot (Linear and Semi-log) (Part 1) | For Cohort A, overlay profiles after the 60mg, 120mg, and overlay profiles on day 1 and day 14 (after 30mg BD) on the same plot For Cohort B, overlay profiles on day 1 and day 14 on the same plot | SAC |
| 4.8. | Systemic PK | PK16a | Individual CCI15106 Plasma Concentration-Time Plot (Linear and Semi-log) (Part 2) | For Cohort B, also overlay profiles on day 1 and day 14 on the same plot (ignore pre-dose PK from day 2 to day 12, and day 15) | SAC |
| 4.9. | Systemic PK | Non-Standard<br>PK_F1 | CCI15106 trough Plasma Concentration versus Study Day (Part 1 and Part 2) | Use line plot, All pre-dose from Day 2 following the BD regimens onwards Linear scale only | SAC |
| 4.10. | Systemic PK | Non-Standard<br>PK_F1 | CCI15106 Plasma Concentration at follow up visit versus Subject ID (Part 1 and Part 2) | Scatter Plot | SAC |
| 4.11. | BAL PK | Non-Standard<br>PK_F2 | Scatter Plot of Lung Drug Concentration versus Subject ID (Part 1 and Part 2) | X Axis: Subject ID<br>Y-Axis: ELF Values | SAC |
| 4.12. | BAL PK | Non-Standard<br>PK_F2 | Scatter Plot of Lung Drug Concentration versus Plasma<br>Drug Concentration (BAL cohorts in Part 1 and Part 2) | data for all patients on same page separate colours for healthy and COPD patients Cohorts B for both parts The template is similar to PK_F2, only change the X-axis to plasma drug concentration. | SAC |

# 11.10.8. ICH Listings

| ICH: Listings | | | | |
|---|---|---|---|---|
| Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| nization | | | | |
| Safety | TA1 | Listing of Randomized and Actual Treatments – Part 1 | This will not include Cohort C, Part 1. | SAC |
| Safety | TA1 | Listing of Randomized and Actual Treatments – Part 2 | | SAC |
| t Disposition | | | | |
| Safety | ES2 | Listing of Reasons for Study Withdrawal – Part 1 | This will not include Cohort C, Part 1. | SAC |
| Safety | ES2 | Listing of Reasons for Study Withdrawal – Part 2 | | SAC |
| Bystander<br>Safety (Part<br>1, Cohort C) | ES2 | Listing of Reasons for Study Withdrawal – Bystander | Only for Cohort C, Part 1. | SAC |
| All<br>Participants<br>Screened | ES7 | Listing of Reasons for Screen Failure – Part 1 | This will not include Cohort C, Part 1. | SAC |
| All<br>Participants<br>Screened | ES7 | Listing of Reasons for Screen Failure – Part 2 | | SAC |
| Bystander<br>Safety (Part<br>1, Cohort C) | ES7 | Listing of Reasons for Screen Failure – Bystander | Only for Cohort C, Part 1. | SAC |
| Safety | SD2 | Listing of Subjects with Study Drug Stopping Record – Part 1 | This will not include Cohort C, Part 1. | SAC |
| Safety | SD2 | Listing of Subjects with Study Drug Stopping Record – Part 2 | | SAC |
| ol Deviations | | | · | , |
| Safety | DV2 | Listing of Important Protocol Deviations – Part 1 | This will not include Cohort C, Part 1. | SAC |
| | Population Safety Safety Disposition Safety Safety Bystander Safety (Part 1, Cohort C) All Participants Screened All Participants Screened Bystander Safety (Part 1, Cohort C) Safety Safety Safety Safety | Population Safety TA1 Safety TA1 Safety TA1 Disposition Safety SD2 Safety SD2 Safety SD2 Safety SD2 Safety SD2 Safety SD2 | Population IDSL / Example Shell Title | Population Pop |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12. | Safety | DV2 | Listing of Important Protocol Deviations – Part 2 | | SAC |
| 13. | Bystander<br>Safety (Part<br>1, Cohort C) | DV2 | Listing of Important Protocol Deviations – Bystander | Only for Cohort C, Part 1. | SAC |
| 14. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 15. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations – Part 2 | | SAC |
| 16. | Bystander<br>Safety (Part<br>1, Cohort C) | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations – Bystander | Only for Cohort C, Part 1. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 17. | Safety | DM2 | Listing of Demographic Characteristics – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 18. | Safety | DM2 | Listing of Demographic Characteristics – Part 2 | | SAC |
| 19. | Bystander<br>Safety (Part<br>1, Cohort C) | DM2 | Listing of Demographic Characteristics – Bystander | Only for Cohort C, Part 1. | SAC |
| 20. | Safety | DM9 | Listing of Race – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 21. | Safety | DM9 | Listing of Race – Part 2 | | SAC |
| 22. | Bystander<br>Safety (Part<br>1, Cohort C) | DM9 | Listing of Race - Bystander | Only for Cohort C, Part 1. | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 23. | Safety | CP_CM3 | Listing of Concomitant Medications – Part 1 | This will not include Cohort C, Part 1. | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Safety | CP_CM3 | Listing of Concomitant Medications – Part 2 | | SAC |
| 25. | Bystander<br>Safety (Part<br>1, Cohort C) | CP_CM3 | Listing of Concomitant Medications – Bystander | Only for Cohort C, Part 1. | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 26. | Safety | EX4 | Listing of Exposure Data – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 27. | Safety | EX4 | Listing of Exposure Data – Part 2 | | SAC |
| 28. | Bystander<br>Safety (Part<br>1, Cohort C) | EX4 | Listing of Exposure Data – Part 2 | | SAC |
| Advers | e Events | | | | |
| 29. | Safety | AE9CP | Listing of All Adverse Events – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 30. | Safety | AE9CP | Listing of All Adverse Events – Part 2 | | SAC |
| 31. | Bystander<br>Safety (Part<br>1, Cohort C) | AE9CP | Listing of All Adverse Events – Bystander | Only for Cohort C, Part 1. | SAC |
| 32. | Safety | AE9CP | Listing of Serious Adverse Events – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 33. | Safety | AE9CP | Listing of Serious Adverse Events – Part 2 | This will not include Cohort C, Part 1. | SAC |
| 34. | Bystander<br>Safety (Part<br>1, Cohort C) | AE9CP | Listing of Serious Adverse Events – Bystander | Only for Cohort C, Part 1. | SAC |
| 35. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Part 1 | This will not include Cohort C, Part 1. | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 36. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Part 2 | | SAC |
| 37. | Bystander<br>Safety (Part<br>1, Cohort C) | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Bystander | Only for Cohort C, Part 1. | SAC |
| All Lab | oratory | | | | |
| 38. | Safety | LB5 | Listing of Haematology Laboratory Data – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 39. | Safety | LB5 | Listing of Haematology Laboratory Data – Part 2 | | SAC |
| 40. | Bystander<br>Safety (Part<br>1, Cohort C) | LB5 | Listing of Haematology Laboratory Data – Bystander | Only for Cohort C, Part 1. | SAC |
| 41. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 42. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data – Part 2 | | SAC |
| 43. | Bystander<br>Safety (Part<br>1, Cohort C) | LB5 | Listing of Clinical Chemistry Laboratory Data – Bystander | Only for Cohort C, Part 1. | SAC |
| 44. | Safety | LB5 | Listing of Coagulation Laboratory Data – Part 1 | This will not include Cohort A and Cohort C, Part 1. | SAC |
| 45. | Safety | LB5 | Listing of Coagulation Laboratory Data – Part 2 | Only for Cohort B, Part 2. | SAC |
| 46. | Safety | UR2a | Listing of Urinalysis Data – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 47. | Safety | UR2a | Listing of Urinalysis Data – Part 2 | | SAC |
| 48. | Bystander<br>Safety (Part<br>1, Cohort C) | UR2a | Listing of Urinalysis Data – Bystander | Only for Cohort C, Part 1. | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 49. | Safety | EG3 | Listing of ECG Values – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 50. | Safety | EG3 | Listing of ECG Values – Part 2 | | SAC |
| 51. | Bystander<br>Safety (Part<br>1, Cohort C) | EG3 | Listing of ECG Values - Bystander | Only for Cohort C, Part 1. | SAC |
| 52. | Safety | EG5 | Listing of ECG Findings – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 53. | Safety | EG5 | Listing of ECG Findings – Part 2 | | SAC |
| 54. | Bystander<br>Safety (Part<br>1, Cohort C) | EG5 | Listing of ECG Findings – Bystander | Only for Cohort C, Part 1. | SAC |
| 55. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Values of Potential Clinical Importance – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 56. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Values of Potential Clinical Importance – Part 2 | | SAC |
| 57. | Bystander<br>Safety (Part<br>1, Cohort C) | EG3 | Listing of All ECG Values for Subjects with Any Values of Potential Clinical Importance – Bystander | Only for Cohort C, Part 1. | SAC |
| Spirom | netry | | | | |
| 58. | Safety | Non-Standard<br>SAFE_L1 | Listing of Spirometry Values – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 59. | Safety | Non-Standard<br>SAFE_L1 | Listing of Spirometry Values – Part 2 | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Teleme | try | | | | |
| 60. | Safety | Non-Standard<br>SAFE_L2 | Listing of Telemetry Values – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 61. | Safety | Non-Standard<br>SAFE_L2 | Listing of Telemetry Values – Part 1 | | SAC |
| Vital Si | gns | | | | |
| 62. | Safety | VS4 | Listing of Vital Signs – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 63. | Safety | VS4 | Listing of Vital Signs – Part 2 | | SAC |
| 64. | Bystander<br>Safety (Part<br>1, Cohort C) | VS4 | Listing of Vital Signs - Bystander | Only for Cohort C, Part 1. | SAC |
| 65. | Safety | VS4 | Listing of All Vital Signs for Subjects with Any values of Potential Clinical Importance – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 66. | Safety | VS4 | Listing of All Vital Signs for Subjects with Any values of Potential Clinical Importance – Part 2 | | SAC |
| 67. | Bystander<br>Safety (Part<br>1, Cohort C) | VS4 | Listing of All Vital Signs for Subjects with Any values of Potential Clinical Importance – Bystander | Only for Cohort C, Part 1. | SAC |

# 11.10.9. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetics | | | | |
| 68. | Systemic PK | PK08 | Listing of CCI15106 Plasma Pharmacokinetic Concentration-<br>Time Data by Cohort and Study Day | | SAC |
| 69. | Systemic PK | PK14 | Listing of Derived CCI15106 Plasma Pharmacokinetic Parameters Cohort and Study Day | | SAC |
| Safety | | | | | |
| 70. | Safety | MH2 | Listing of Medical Conditions – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 71. | Safety | MH2 | Listing of Medical Conditions – Part 2 | | SAC |
| 72. | Bystander<br>Safety (Part<br>1, Cohort C) | MH2 | Listing of Medical Conditions – Bystander | Only for Cohort C, Part 1. | SAC |
| 73. | Safety | SU2 | Listing of Substance Use – Part 1 | This will not include Cohort C, Part 1. | SAC |
| 74. | Safety | SU2 | Listing of Substance Use – Part 2 | | SAC |
| 75. | Bystander<br>Safety (Part<br>1, Cohort C) | SU2 | Listing of Substance Use – Bystander | Only for Cohort C, Part 1. | SAC |
| 76. | All Screened<br>Population | IE4 | Listing of Study Eligibility – Part 1 | | SAC |
| 77. | All Screened<br>Population | IE4 | Listing of Study Eligibility – Part 2 | | SAC |

205822

## 11.11. Appendix 11: Example Mock Shells for Data Displays

Example SAFE\_T1
Protocol: 205822
Population: Safety

Page 1 of 2

Table 1.61
Summary of Demographic Characteristics - Part 1

| | | Cohort B (N=12) | Placebo<br>(N=4) |
|---|---|---|---|
| Sex | | | |
| n | 6 | 12 | 4 |
| Male | 6 (100%) | 12 (100%) | 4 (100%) |
| Female | 0 | 0 | 0 |
| Age (y) | | | |
| n | 6 | 12 | 4 |
| Mean | 39.8 | 35.4 | 43.3 |
| SD | 9.75 | 11.18 | 9.54 |
| Median | 40.0 | 31.0 | 44.0 |
| Min. | 25 | 25 | 32 |
| Max. | 52 | 57 | 53 |
| Ethnicity | | | |
| n | 6 | 12 | 4 |
| HISPANIC OR LATINO | 0 | 1 (8%) | 0 |
| NOT HISPANIC OR LATINO | 6 (100%) | 11 (92%) | 4 (100%) |
| Race | | | |
| n | 6 | 12 | 4 |
| WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 5 (83%) | 9 (75%) | 4 (100%) |
| AFRICAN AMERICAN/AFRICAN HERITAGE | 1 (17%) | 2 (17%) | 0 |
| Multiple . | 0 | 1 (8%) | 0 |

.

Example SAFE\_T2
Protocol: 205822

Population: Safety

Table X
Summary of Telemetry Findings - Part 1

| | _ | | | ohort B<br>(N=160) | Placebo (N=160) | |
|---|---|---|---|---|---|---|
| Time Period 1 | | | | | | |
| n | 156 | | 160 | | 160 | |
| Normal | 81 | (52%) | 90 | (56%) | 90 | (56%) |
| Abnormal, not clinically significant | 75 | (48%) | 69 | (43%) | 69 | (43%) |
| Abnormal, clinically significant | 0 | | 1 | (<1%) | 1 | (<1%) |
| Time Period 2 | | | | | | |
| n | 117 | | 123 | | 123 | |
| Normal | 50 | (43%) | 67 | (54%) | 67 | (54%) |
| Abnormal, not clinically significant | 64 | (55%) | 55 | (45%) | 55 | (45%) |
| Abnormal, clinically significant | 2 | (2%) | 1 | (<1%) | 1 | (<1%) |

•

.

.

Example SAFE\_T3
Protocol: 205822

Population: Safety

Table X Summary of Spirometry Results - Part 1

| | CCI15106 | CCI15106 | CCI15106 | Placebo |
|-----------------|----------|----------|----------|---------|
| | 60mg SD | 120mg SD | 30mg BID | |
| | (N=157) | (N=160) | (N=160) | (N=160) |
| Time Period 1 | | | | |
| n | 156 | 160 | | 160 |
| %Predicted FEV1 | 52% | 56% | | 56% |
| %Predicted FVC | 55% | 45% | | 45% |
| Time Period 2 | | | | |
| n | 117 | 123 | | 123 |
| %Predicted FEV1 | 52% | 56% | | 56% |
| %Predicted FVC | 55% | 45% | | 45% |
| • | | | | |
| • | | | | |
| • | | | | |
| • | | | | |

<sup>%</sup> Predicted FEV1 = (Max FEV1/Predicted Normal FEV1)x100

<sup>%</sup> Predicted FVC = (Max FVC/Predicted Normal FVC)x100

Example SAFE\_T4
Protocol: 205822
Population: Safety

Page 1 of 2

Table 3.51
Summary of All Serious Adverse Events - Part1

| System Organ Class Preferred Term | | CCI15106<br>120 mg SD | | CCI15106<br>60 mg BID | Placebo |
|---|---|---|---|---|---|
| ANY EVENT | 1 (17%) | 0 | 4 (67%) | 9 (75%) | 1 (25%) |
| Blood and lymphatic system disorders | | | | | |
| Any event | 0 | 0 | 0 | 1 (8%) | 0 |
| Lymphadenopathy | 0 | 0 | 0 | 1 (8%) | 0 |
| Gastrointestinal disorders | | | | | |
| Any event | 0 | 0 | 1 (17%) | 2 (17%) | 0 |
| Diarrhoea | 0 | 0 | 0 | 1 (8%) | 0 |
| Mouth ulceration | 0 | 0 | 1 (17%) | 0 | 0 |
| Vomiting | 0 | 0 | 0 | 2 (17%) | 0 |
| General disorders and administration | | | | | |
| site conditions | | | | | |
| Any event | 0 | 0 | 0 | 5 (42%) | 0 |
| Asthenia | 0 | 0 | 0 | 1 (8%) | 0 |
| Chest pain | 0 | 0 | 0 | 1 (8%) | 0 |
| Feeling hot | 0 | 0 | 0 | 2 (17%) | 0 |
| Influenza like illness | 0 | 0 | 0 | 1 (8%) | 0 |
| Malaise | 0 | 0 | 0 | 3 (25%) | 0 |
| Infections and infestations | | | | | |
| Any event | 0 | 0 | 1 (17%) | 1 (8%) | 0 |
| Nasopharyngitis | 0 | 0 | 1 (17%) | 0 | 0 |
| Upper respiratory tract infection | 0 | 0 | 0 | 1 (8%) | 0 |
| Injury, poisoning and procedural | | | | | |

Injury, poisoning and procedural
complications

.

Example SAFE\_T5
Protocol: 205822

Protocol: 205822 
Population: Safety

Table X
Summary of Extent of Exposure to Study Treatment - Part 1

| | Period | | 60mg(HV) | CCI15106 SD<br>120mg(HV)<br>(N=6) | 30mg(HV) | | Placebo(HV)<br>(N=4) |
|---|---|---|---|---|---|---|---|
| Time on Study Treatment (days) [1] | PERIOD 1 | n | х | Х | Х | XX | Х |
| | | Mean | X.X | X | X | XX.X | XX.X |
| | | SD | X.XX | X | X | X.XX | XX.XX |
| | | Median | X • X | X | X | XX.X | XX.X |
| | | Min. | X | X | X | XX | X |
| | | Max. | X | X | X | XX | XX |
| | PERIOD 2 | n | X | X | X | X | X |
| | | Mean | X | X . X | X | X | X . X |
| | | SD | X | X.XX | X | X | X.XX |
| | | Median | X | X . X | X | X | X . X |
| | | Min. | X | X | X | X | X |
| | | Max. | X | X | X | X | X |
| | PERIOD 3 | n | X | X | X | X | X |
| | | Mean | X | X | XX.X | X | XX.X |
| | | SD | X | X | X.XX | X | X.XX |
| | | Median | X | X | XX.X | X | XX.X |
| | | Min. | X | X | XX | X | XX |
| | | Max. | X | Х | XX | Х | XX |
| Subject Daily Dose (mg) [2] | PERIOD 1 | n | X | Х | X | XX | X |
| | | Mean | XX.X | X | X | XX.X | X.X |
| | | SD | X.XX | Х | X | X.XX | X.XX |

| | | Median | XX.X | X | X | XX.X | X . X |
|---|---|---|---|---|---|---|---|
| | | Min. | XX | X | X | XX | X |
| | | Max. | XX | X | X | XX | X |
| | PERIOD 2 | n | X | X | X | X | X |
| | | Mean | X | XX.X | X | X | X . X |
| | | SD | X | X.XX | X | X | X.XX |
| | | Median | X | XX.X | X | X | X . X |
| | | Min. | X | X | X | X | X |
| | | Max. | X | XX | X | X | X |
| | PERIOD 3 | n | X | X | X | X | X |
| | | Mean | X | X | XX.X | X | X . X |
| | | SD | X | X | X.XX | X | X.XX |
| | | Median | X | X | X . X | X | x.x |
| | | Min. | X | X | XX | X | Х |
| | Max. | Х | Х | XX | Х | X | |
| Cumulative Actual Dose (mg) | PERIOD 1 | n | Х | X | X | XX | X |
| | | Mean | XX.X | X | X | X.X | X . X |
| | | SD | X.XX | X | X | X.XX | X.XX |
| | | Median | XX.X | X | X | X.X | X.X |
| | | Min. | X | X | X | XX | Х |
| | | Max. | XX | X | X | XX | X |
| | PERIOD 2 | n | Х | X | X | X | X |
| | | Mean | Х | X . X | X | X | x.x |
| | | SD | Х | X.XX | X | Х | X.XX |
| | | Median | Х | X . X | X | Х | x.x |
| | | Min. | X | XX | Х | Х | Х |
| | | Max. | Х | XX | X | Х | Х |
| | PERIOD 3 | n | Х | X | X | X | Х |
| | | Mean | Х | X | XX.X | X | x.x |
| | | SD | X | X | X . X | X | X.XX |
| | | Median | X | X | XX.X | X | x.x |
| | | Min. | X | X | XX | X | X |
| | | Max. | X | X | XX | X | X |

205822

Note: [1] The time on study drug does not exclude dose interruptions.
[2] The subject daily dose (the cumulative actual dose divide by the duration of exposure) is calculated for each subject first and the summary statistics are calculated based on the subject average daily dose.

205822


Example SAFE\_T6
Protocol: 205822

Population: Safety

Table X
Frequency of Worst Change from Baseline Values of QTcB and QTcF by PCI Category

| ECG Test | Visit | Category | Placebo (N=12) | CCI15106-CFI -<br>1 capsule -<br>Single Dose<br>(N=6) | |
|---|---|---|---|---|---|
| QTcB Interval, Aggregate (msec) | BASELINE | n | 12 | 6 | 6 |
| | Worst Post<br>Baseline | n<br>Increase<=30<br>30 <increase<=60<br>Increase&gt;60</increase<=60<br> | 12<br>12(100%)<br>0 | 6<br>6(100%)<br>0 | 6<br>6(100%)<br>0 |
| QTcF Interval,<br>Aggregate (msec) | Baseline | n | 12 | 6 | 6 |
| | Worst Post<br>Baseline | n Increase<=30 30 <increase<=60 increase="">60</increase<=60> | 12<br>12(100%)<br>0 | 6<br>6(100%)<br>0 | 6<br>6(100%)<br>0 |

Example SAFE\_T7
Protocol: 205822
Population: Safety

rotocol: 205822 

Table X
Frequency of Maximum ECG Values by PCI Category

| ECG Test | Visit | Category | Placebo<br>(N=12) | 1 capsule -<br>Single Dose | Single Dose |
|---|---|---|---|---|---|
| PR Interval, Aggregate (msec) | BASELINE | n | 12 | 6 | 6 |
| nggregate (mete) | | Value<110<br>110<=Value<=220<br>Value>220 | | 0<br>6(100%)<br>0 | 0<br>6(100%)<br>0 |
| | WORST POST<br>BASELINE | n<br>Value<110<br>110<=Value<=220<br>Value>220 | - | 6<br>0<br>6(100%)<br>0 | 6<br>0<br>6(100%)<br>0 |
| QRS Duration,<br>Aggregate (msec) | SCREENING | n | 12 | 6 | 6 |
| 1199209000 (111000) | | Value<75<br>75<=Value<=110<br>Value>110 | , , | 0<br>6 (100%)<br>0 | 0<br>6(100%)<br>0 |
| | WORST POST<br>BASELINE | n<br>Value<75<br>75<=Value<=110<br>Value>110 | 12<br>0<br>11 (92%)<br>1 (8%) | 6<br>0<br>6(100%)<br>0 | 6<br>0<br>6(100%)<br>0 |
| QTcB Interval,<br>Aggregate (msec) | SCREENING | n | 12 | 6 | 6 |

205822

| | Value<=450<br>450 <value<480< th=""><th>11 (92%)<br/>1 (8%)</th><th>6 (100%)<br/>0</th><th>6 (100%)<br/>0</th></value<480<> | 11 (92%)<br>1 (8%) | 6 (100%)<br>0 | 6 (100%)<br>0 |
|---|---|---|---|---|
| | 480<=Value<500 | 0 | 0 | 0 |
| | Value>=500 | 0 | 0 | 0 |
| WORST POST | n | 12 | 6 | 6 |
| BASELINE | Value<=450 | 11 (92%) | 5 (83%) | 6 (100%) |
| | 450 <value<480< td=""><td>1 (8%)</td><td>1 (17%)</td><td>0</td></value<480<> | 1 (8%) | 1 (17%) | 0 |
| | 480<=Value<500 | 0 | 0 | 0 |
| | Value>=500 | 0 | 0 | 0 |

Repeat for QTcF

Note: Percentages may not add up to 100 for QRS Duration and PR Interval as there is a possibility of a patient being counted under both low and high categories.

205822

Example : PK\_T1 Page 1 of n : 205822

Population : Systemic PK

Table 3.1.13
Summary of Assessment of Dose Proportionality (Part 1 and Part 2)

| | | | Slope | | | _ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | Study | n | Estimate | SE | 90% CI | Estimate | SE | 90% CI | Coefficient of |
| | Day | | | | | | | | Determination |

Note(s): CI = confidence interval; SE = standard error.

Source: SAS Output XX

205822

Example : PK\_T2 Page 1 of n

Protocol : 205822 Population : Systemic PK

Table 3.1.16 Summary of Assessment of Steady State (Part 1 and Part 2)

| | | | Slope | Slope |
|-----------|---|----------|-------|--------|
| Parameter | n | Estimate | SE | 90% CI |

Note(s): CI = confidence interval; SE = standard error.

Source: SAS Output XX

CONFIDENTIAL 205822

Example : PK\_T3 Page 1 of n
Protocol : 205822

Population : Systemic PK

Table 3.1.17
Summary of Assessment of Accumulation (Part 1 and Part 2)

| | | | | | Geometric | Ratio of | | |
|---|---|---|---|---|---|---|---|---|
| Dose | Parameter | Study | | Geometric | LS Mean | Geometric | | |
| Level | (unit) | Day | n | LS Mean | 95% CI | Means | 90% CI | p-value |

Note(s): LS = least squares; CI = confidence interval.

Accumulation was assessed using a linear mixed effects model with day as a fixed effect and subject as a random effect.

205822

Source: SAS Output XX

Example : SAFE\_L1 Page 1 of n

Protocol : 205822

Population : Safety (Part 1)

Listing 59
Listing of Spirometry Values – Part 1

| | | | | | | | Spirometry | 7 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Time | | | | | | | |
| | Visit | | | of | | | | | | | |
| Cohort | / | | | first | | | | | | | |
| / | Study | Visit | | exhal | | | | | | Highest | |
| Subj. | Day | date | Test | ation | Reading | 1 | Reading 2 | Reading 3 | 3 | reading | %predicted |

205822

Source: SAS Output XX

Example : SAFE\_L2 Page 1 of n

Protocol : 205822

Population : Safety (Part 1)

Listing 62
Listing of Telemetry Values – Part 1

| Cohort | Visit<br>/ | | | | | | |
|---|---|---|---|---|---|---|---|
| / | _ | Visit | | Time | Date | Time | |
| Subj. | Day | date | started | started | stopped | stopped | Telemetry Result |

Example : PK\_F1

Protocol : 205822 Population : Systemic PK

Figure xxx: CCI15106 trough Plasma Concentration versus Study Day (Part 2)



Example : PK\_F2

Protocol : 205822 Population : BAL PK

Figure XXX Scatter Plot of Lung Drug Concentration versus Subject ID (Part 1 and Part 2)

